CLINICAL TRIAL: NCT01207570
Title: Effect of Endermotherapy on Passive Ankle Range of Motion in Children With Developmental Disabilities
Brief Title: Endermotherapy for Children With Developmental Disabilities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Phoelia Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20091207001
Record Dates: First submitted 2010-09-17; First posted 2010-09-23 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Cerebral Palsy; Developmental Delay
Keywords: flexibility; muscle; stretching; cerebral palsy; developmental
MeSH Terms: conditions — Cerebral Palsy; Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endermotherapy (Experimental): The subjects in the experimental group will receive a single session (5 minutes) of endermotherapy) applied to the gastrocnemius/soleus muscle group in the more affected side. The treatment will b e carried out by a qualified physiotherapist.
  Interventions: Procedure: Endermotherapy
- Passive stretching (Active Comparator): The subjects in this group will receive a single session of passive stretching of the gastrocnemius/soleus muscle for 5 minutes.
  Interventions: Procedure: Passive manual stretching

INTERVENTIONS:
Procedure: Endermotherapy — The subjects will receive a single session of endermotherapy applied to the gastrocnemius/soleus muscle on the more affected side for 5 minutes. The treatment will be conducted by a qualified physiotherapist.
  Arms: Endermotherapy
Procedure: Passive manual stretching — The subjects will receive a single session of passive manual stretching of the gastrocnemius/soleus muscle on the more affected side. The treatment will be given by a qualified physiotherapist.
  Arms: Passive stretching

SUMMARY:
Children with developmental disabilities often sustain decreased range of motion in their extremities. The decrease in flexibility may be due to neuromuscular disorders such as spasticity or dystonia. Other causes may be imbalance in muscle strength surrounding a joint, leading to inappropriate habitual posture. Over time, muscle contracture may result for those muscle groups that are placed in a shortened position for an extended period of time. The most common site of muscle contractures among these children are gastrocnemius/soleus (lower limbs), and latissimus dorsi muscles (upper limbs). Muscle contractures can lead to further decline in functional abilities. Therefore, it is important to identify effective intervention strategies to enhance or maintain muscle flexibility in children with developmental dysfunctions.

Commercially available endermotherapy device has been used to soften scar tissue following burn injuries. The mechanical stimulation applied may also have beneficial effects on relaxing the muscle tissue. The overall aim of the proposed study is to determine whether endermotherapy treatment has immediate effect in improving joint range of motion among children with developmental disabilities.

The research hypothesis is that children in the endermotherapy group will have significantly more gain in ankle passive range of motion than those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 2 and 6.
* children with diagnosis of cerebral palsy or developmental disabilities.
* Has limited ankle dorsiflexion range of motion (less than 20 degrees)

Exclusion Criteria:

* Other serious illnesses that preclude participation

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Y P, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Heep Hong Society, Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited from Heep Hong Society, a non-governmental organization that provides rehabilitation services for children with disabilities.
  The recruitment period was between January 2010 and June 2010.
Pre-assignment Details: No significant events.
Period: The First Stage (Before Crossover)
Arm/Group | Endermotherapy | Passive Stretching
Started | 23 | 31
Completed | 23 | 31
Not Completed | 0 | 0
Period: The Second Stage (After Crossover)
Arm/Group | Endermotherapy | Passive Stretching
Started | 31 | 23
Completed | 31 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endermotherapy | Passive Stretching | Total
Number analyzed (Participants) | 23 | 31 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 31 | 54
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 4.7 (1.5) | 4.9 (1.2) | 4.8 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 15 | 22
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  Hong Kong | 23 | 31 | 54

OUTCOME MEASURES:

1. Primary Outcome: Ankle Passive Range of Motion
Description: The ankle passive range of motion will be measured by a Myrin goniometer.
Time Frame: day 1 before treatment
Population: All subjects received the intended treatment protocol and were included in the analysis. ITT was used to analyze the data.
Measure: Mean (Standard Deviation); unit: degree
Groups:
- Endermotherapy: A single endermotherapy treatment session
- Passive Stretching: A single passive stretching session
Arm/Group | Endermotherapy | Passive Stretching
Number analyzed (Participants) | 23 | 31
degree | 8.3 (8.1) | 10.4 (6.0)

2. Primary Outcome: Ankle Passive Range of Motion
Description: Ankle passive range of motion at day 4 before the crossover treatment
Time Frame: day 4 before treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree
Groups:
- Endermotherapy: A single session of endermotherapy treatment
- Passive Stretching: A single session of passive stretching
Arm/Group | Endermotherapy | Passive Stretching
Number analyzed (Participants) | 31 | 23
degree | 11.6 (6.0) | 11.3 (8.3)

3. Primary Outcome: Ankle Passive Range of Motion
Description: Ankle dorsiflexion passive range of motion
Time Frame: Day 1 after treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Endermotherapy | Passive Stretching
Number analyzed (Participants) | 23 | 31
degree | 12.2 (8.6) | 14.9 (6.7)

4. Primary Outcome: Ankle Passive Range of Motion
Description: Ankle passive range of motion on day 4 after the crossover treatment
Time Frame: Day 4 after treatment
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Endermotherapy | Passive Stretching
Number analyzed (Participants) | 23 | 31
degree | 15.9 (6.7) | 13.5 (8.4)

ADVERSE EVENTS:
Arm/Group | Endermotherapy | Passive Stretching
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No